CLINICAL TRIAL: NCT06793813
Title: A Phase II Trial of Cadonilimab (PD-1/CTLA-4 Bispecific Antibody) in Combination with Bevacizumab and Docetaxel in Patients (pts) with Checkpoint Inhibitor (CPI)-experienced Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: Cadonilimab in Patients (Pts) with Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jie Wang, Chief Physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-017
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-01

CONDITIONS: Stage IVB Lung Cancer; Non-Squamous
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm A (cadonilimab，bevacizumab，docetaxel ) (Experimental)
  Interventions: Drug: cadonilimab，bevacizumab，docetaxel

INTERVENTIONS:
Drug: cadonilimab，bevacizumab，docetaxel — Patients receive Cadonilimab IV over 90 minutes on day 1. Patients also receive bevacizumab 7.5mg/kg IV on day 1 and docetaxel 60-75 mg/m2 IV over 60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

SUMMARY:
This phase II trial studies how well cadonilimab combined with Bevacizumab and docetaxel work in treating patients with non-squamous and stage IV non-small cell lung cancer. Cadonilimab, a PD-1/CTLA-4 bispecific antibody, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Bevacizumab can regulate tumor microenvironment. Docetaxel was used in standard of care chemotherapy for non-small cell lung cancer, work to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving cadonilimab, bevacizumab and docetaxel together may work better in treating patients with non-squamous non-small lung cancer compared to standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old
2. Locally advanced (stage IIIB/IIIC) that cannot be resected by radical surgery and cannot accept radical synchronous/sequential radiotherapy and chemotherapy and metastatic (stage IV) non-squamous NSCLC confirmed by histology or cytology
3. Patients must have progressed on at most a PD-1/L1 inhibitor and a platinum-based chemotherapy (combined or sequential, regardless of sequence), and at least two cycles of PD-1/L1 inhibitor (combined or non-combined chemotherapy) with clinical benefits (PFS ≥ 3 months)
4. Patients must not have EGFR sensitizing mutations, EGFR T790M mutation, ALK gene fusion, and ROS 1 gene rearrangement, and BRAF V600E mutation.
5. Has measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
6. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
7. Life expectancy > 12 weeks as determined by the investigator
8. Patients must have at least one measurable lesion (as defined by RECIST v1.1), which is suitable for repeated and accurate measurement
9. Absolute neutrophil count (ANC) ≥ 1500/uL (collected within 10 days prior to the start of study treatment)
10. Platelets ≥ 100 000/uL (collected within 10 days prior to the start of study treatment)
11. Hemoglobin ≥ 9.0 g/dL (collected within 10 days prior to the start of study treatment)
12. Creatinine clearance [CrCl]) ≥ 50 mL/min(Creatinine clearance (CrCl) should be calculated per institutional standard)
13. Total bilirubin ≤ 1.5 x ULN (collected within 10 days prior to the start of study treatment)
14. Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 x ULN (≤ 5 x ULN for participants with liver metastases) (collected within 10 days prior to the start of study treatment
15. Serum albumin(ALB)≥28 g/L
16. International standardized ratio (INR) and activated partial thrombin time (APTT) ≤ 1.5 × ULN
17. Left ventricular ejection fraction (LVEF) ≥ 50%
18. A male participant must agree to use a contraception during the treatment period plus an additional 120 days after the last dose of study treatment and refrain from donating sperm during this period
19. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP) OR
    2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days plus 30 days (a menstruation cycle) after the last dose of study treatment

Exclusion Criteria:

1. Previously received treatment for tumor immune mechanism other than any anti-PD-1/L1 inhibitor for advanced NSCLC stage, such as CTLA-4（CD152）、TIGIT、OX-40、CD137、ICOS、CD40、CD47、CD73、GITR、TOX、LAG-3、TIM3、SIRPα、BTLA（CD272）、VISTA（B7-H5）、LIGHT（CD258）、B7-H3（CD276）、 B7-H4（VTCN1）、HVEM、CD80/CD86、MHC Ⅱ、GAL9、IDO、PVR（CD155）、Nectin-2（CD112）.
2. Patients have prior exposure to docetaxel, bevacizumab
3. The last systemic anti-tumor treatment (chemotherapy, immunotherapy, biological agents, anti-angiogenic drugs, etc.) was received within 3 weeks before the first administration.
4. The following treatments were received within 2 weeks before the first administration: TKI treatment, hormone anti-tumor treatment, palliative local treatment for non-target lesions Non-specific immunomodulatory therapy (such as interleukin, interferon, thymosin, tumor necrosis factor, etc., excluding IL-11 for thrombocytopenia).
5. Patients with explosive progress.
6. Patients with other active malignant tumors except for NSCLC within 3 years before enrollment. Patients with other malignant tumors that have been cured by local treatment, such as basal or cutaneous squamous cell carcinoma, superficial bladder cancer cancer, cervical or breast cancer in situ, are not excluded.
7. Patients with active autoimmune diseases that require systemic treatment in the past two years (such as the use of disease improvement drugs, corticosteroids, immunosuppressants) (excluding irAE caused by the use of PD-1/L1 inhibitors). Replacement therapy (such as thyroid hormone, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered as a systemic treatment.
8. Patients can not swallow pills, with malabsorption syndrome, or any condition that affects gastrointestinal absorption;
9. Patients with active or previous history of inflammatory bowel disease (such as Crohn's disease, ulcerative colitis or chronic diarrhea).
10. Patients have a history of immune deficiency, with HIV antibody test positive or use systemic corticosteroids or other immunosuppressants for a long time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
6-month progression-free survival | up to 6 months
  Will be determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Will be reported and its 95% confidence intervals will be estimated using the Clopper-Pearson method. PFS rates of two patient groups stratified by binary biomarker (PD-L1 and KRAS status), respectively will be estimated with the Kaplan-Meier method and compared using the log-rank test, respectively. Cox proportional hazards models will be further used in the multivariable analyses to assess adjusted effect of PD-L1 and KRAS status on the patients' PFS after adjusting for other factors. Interaction terms between these factors will also be tested for statistical significance. The proportional hazards assumption will be evaluated graphically and analytically with regression diagnostics. Violations of the proportional hazards assumptions will be addressed by use of time-dependent covariates or extended Cox regression models.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided